CLINICAL TRIAL: NCT01000883
Title: Correlation of Molecular Markers With Response to Therapy and Breast Cancer Behavior
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 9819; P50CA058223 (NIH); P30CA016086 (NIH); 05-2015 Also (05-MED-521-ORC) (Other: IRB assigned number)
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary tumor and metastatic site tumor tissue; whole blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: biologic sample preservation procedure — approximately 16-20 milligrams of tumor tissue per core will be obtained for research purposes.
Other: laboratory biomarker analysis — Evaluation of biomarkers will occur as questions are asked in subsequent correlative studies.
Procedure: biopsy — cancer tissue will be taken from the primary breast cancer site as well as the metastatic tumor sites. Two tubes of whole blood will also be collected.

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tissue and blood samples from women with locally advanced or metastatic breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

* Collect , catalogue, and store biological specimens from patients with locally advanced or metastatic breast cancer
* To collect clinical data from these patients containing identifiers, demographics, epidemiologic review, clinical evaluation, treatment, and long-term follow-up.
* To provide an efficient bi-directional flow of clinical information and specimens between laboratory and clinical scientists in order to foster innovative translational research.

OUTLINE: This is a multicenter study.

Patients undergo core biopsy and blood sampling at diagnosis, between chemotherapy regimens, and prior to definitive surgery. Tumor markers are assessed using immunohistochemistry and flow cytometry.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

High suspicion of or known breast cancer (early or metastatic)

Lesion accessible for safe biopsy (as deemed by the treating physician).

Age ≥ 18 years.

ECOG performance status 0 - 2.

Ability to understand and willingness to sign an informed consent document.

If receiving therapeutic anticoagulation; it should be discontinued temporarily prior to biopsy for a length of time to be determined by the study doctor.

Adequate marrow function, defined as absolute neutrophil count ≥ 1.5 x 109/L and platelets ≥ 100 x 109/L required only for biopsies of vital organs (lung, liver, etc.)

Exclusion Criteria:

Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety.

Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

History of serious or life-threatening allergic reaction to local anesthetics (i.e. lidocaine, xylocaine)

Pregnant women are excluded because there may be an increased risk to both mother and fetus in the setting of conscious sedation, which is required for biopsies of certain anatomic sites (e.g. liver, lung). Also, ionizing radiation from CT-guided biopsies may pose a risk to the unborn fetus.

Cardiac disease making it unsafe to biopsy in the opinion of the treating physician.

If patients receiving bevacizumab or other angiogenesis inhibitors are less than 6 weeks from last dose of the angiogenesis inhibitor, they should not undergo research core biopsies of vital organs (lung, liver, etc.) on this protocol because of the concern for the possibility of increased bleeding risk and delayed healing. Patients receiving bevacizumab or other angiogenesis inhibitors who are undergoing a research biopsy of the breast, peripheral lymph node or a skin punch biopsy must be two weeks from the last dose of the angiogenesis inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from those individuals receiving diagnostic and treatment related biopsies at the University of North Carolina at Chapel Hill.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1998-12-01 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Generation of a biorepository for current and future correlative research studies | Diagnosis, between treatments,7-14 days after start of treatment and at time of definitive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: web address for Lineberger Comprehensive Cancer Center at UNC — http://unclineberger.org
- See also: web address for the National Cancer Institute — http://www.cancer.gov